CLINICAL TRIAL: NCT05320523
Title: Simultaneous Deep Brain Stimulation of the Globus Pallidus Internus and the Nucleus Basalis of Meynert in Patients With Parkinson's Disease and Mild Cognitive Impairment
Brief Title: Simultaneous DBS of the GPi and the NBM in Patients With Parkinson's Disease and Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 38865720.1.0000.0068
Record Dates: First submitted 2022-03-14; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment
Keywords: Parkinson's disease; Mild cognitive impairment; Globus Pallidus internus (GPi) Stimulation; Nucleus basalis of Meynert (NBM) Stimulation; Deep Brain Stimulation (DBS)
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- GPi stimulation + NBM stimulation (Active Comparator): effective neurostimulation of the Nucleus basalis Meynert combined with globus pallidus internus (GPi) stimulation using Vercise deep brain stimulation
  Interventions: Device: Deep brain stimulation implantation of a Vercise neurostimulation system in GPi and NBM.; Device: GPi stimulation; Device: NBM stimulation
- GPi stimulation + sham stimulation (Sham Comparator): ineffective neurostimulation of the Nucleus basalis Meynert combined with subthalamic nucleus (STN) stimulation using Vercise deep brain stimulation
  Interventions: Device: Deep brain stimulation implantation of a Vercise neurostimulation system in GPi and NBM.; Device: GPi stimulation; Device: Sham stimulation

INTERVENTIONS:
Device: Deep brain stimulation implantation of a Vercise neurostimulation system in GPi and NBM. — Deep brain stimulation implantation of a Vercise neurostimulation system in GPi and NBM, at the same trajectory.
Device: GPi stimulation — Bilateral high-frequency neurostimulation of the GPi using a Vercise neurostimulation system
Device: NBM stimulation — Bilateral low-frequency neurostimulation of the NBM using a Vercise neurostimulation system
  Arms: GPi stimulation + NBM stimulation
Device: Sham stimulation — Ineffective neurostimulation by setting 0mA output at the Vercise neurostimulation system
  Arms: GPi stimulation + sham stimulation

SUMMARY:
Phase 1 study evaluating the safety of combined bilateral globus pallidus internus (GPi) and nucleus basalis of Meynert (NBM) stimulation in treating levodopa responsive motor symptoms of Parkinsonism and cognitive dysfunction, respectively, in patients with moderate to advanced Parkinson's disease having mild cognitive impairment.

DETAILED DESCRIPTION:
This study aims to provide a proof of safety of combined bilateral Globus Pallidus internus (GPi) and Nucleus Basalis of Meynert (NBM) stimulation in patients with moderate to advanced Parkinson's disease having mild cognitive impairment.

GPi stimulation with high-frequency ameliorates the cardinal motor symptoms and motor complications in Parkinson's disease patients, and this present study also wants to determine if additional NBM stimulation, with low-frequency stimulation, improves or slows progression of cognitive decline in patients with moderate to advanced Parkinson's disease having mild cognitive impairment, and to evaluate the effect of NBM stimulation on gait and balance impairment.

Study Design: Prospective single center Phase 1 study with double-blind randomized delayed activation of basal nucleus of Meynert neurostimulation (staggered onset design).

Planned Number of Subjects: 10 patients.

Planned Number of Sites / Countries: Single center in Brazil.

Study schedule:

* Presurgical baseline evaluation (motor on and off medication state; cognitive testing in best motor on state).
* DBS Implant Procedure.
* Postsurgical baseline evaluation (motor off state; cognitive testing in best motor on state) at 3±1 weeks after surgery and activation of globus pallidus internus neurostimulation using individualized stimulation parameters after a standard monopolar review.
* Regular adjustments of the GPi stimulation parameters aiming at the best motor improvement.
* Visit 1 (16 weeks after activation of GPi neurostimulation): motor off medication + GPi stimulation state, cognitive testing in on medication + GPi stimulation state. Randomization and blinded activation of NBM neurostimulation according to a 1:1 scheme.
* Visit 2 (16 weeks after randomization): motor off and on medication + stimulation state (GPi stimulation ± NBM stimulation); cognitive testing in motor on medication + stimulation state (GPi stimulation ± NBM stimulation). Activation of NBM neurostimulation in all patients.
* Visit 3 (16 weeks after activation of NBM stimulation in all patients): motor off and on medication + GPi and NBM stimulation state; cognitive testing in motor on medication + GPi and NBM stimulation state.
* Annual follow-up visit for up to 5 years after activation of NBM stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age at the time of enrollment: 50 - 75 years.
* Diagnosis of idiopathic PD according to Movement Disorders Society (MDS) criteria (Albanese et al., 2017).
* Mild cognitive impairment (MCI) related to Parkinson's disease according to MDS criteria. (Livtan et al. 2012).
* Duration of bilateral idiopathic PD: ≥ 5 years of motor symptoms.
* Modified Hoehn and Yahr stage ≥ 2 on off medication state.
* UPDRS subset III (motor) ≥ 30 points on off medication state.
* Levodopa must improve PD symptoms by ≥ 30% in a levodopa challenge test, as measured by UPDRS subset III score.
* Presence of motor complications related to Parkinson's disease.
* Be willing and able to comply with all visits and study related procedures
* Able to understand the study requirements and the treatment procedures and to provide written informed consent before any study-specific tests or procedures are performed.

Exclusion Criteria:

* Alcohol or drug abuse.
* Any significant psychiatric problems, including acute confusional state (delirium), ongoing psychosis, or clinically significant depression.
* Contraindications for deep brain stimulation (DBS) surgery.
* Heart failure, heart disease or any condition that contraindicates surgical procedures.
* Pacemaker or other active implanted stimulators.
* Clearly established Parkinson's disease dementia according to Movement Disorders Criteria.
* Participation in another drug, device, or biologics trial concurrently.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Safety of combined bilateral Globus Pallidus internus (GPi) and Nucleus Basalis of Meynert (NBM) stimulation in patients with moderate to advanced Parkinson's disease with mild cognitive impairment as determined by reported adverse events. | 36 weeks
  Safety of combined bilateral GPi and NBM stimulation in patients with moderate to advanced Parkinson's disease having mild cognitive impairment as determined by reported adverse events.

SECONDARY OUTCOMES:
Change in Parkinson's Disease - Cognitive Rating Scale (PD-CRS). | 36 weeks
  This scale can range from 0 to 134, and higher scores mean a better outcome.
Change in Mattis Dementia Rating Scale. | 36 weeks
  This scale can range from 0 to 144, and higher scores mean a better outcome.
Change in Verbal Fluency Battery. | 36 weeks
  FAS and animals
Change in Trail Making Task. | 36 weeks
  Trail Making Task Part A + B.
Change in Stroop Test. | 36 weeks
  Stroop Test (Victoria Version).
Change in Symbol Digit Modalities Test. | 36 weeks
  Digit symbol coding - WAIS.
Change in Parkinson's Disease Questionnaire for quality of life (PDQ-39). | 36 weeks
  This questionnaire can range from 0 to 100%, and higher scores mean a worse outcome.
Change in Questionnaire of the EuroQol-group (EQ-5D-5L). | 36 weeks
  This questionnaire can range from 0 to 25, and higher scores mean a worse outcome.
Change in Unified Parkinson's Disease Rating Scale section I (UPDRS I). | 36 weeks
  This scale can range from 0 to 52, and higher scores mean a worse outcome.
Change in Unified Parkinson's Disease Rating Scale section II (UPDRS II). | 36 weeks
  This scale can range from 0 to 52, and higher scores mean a worse outcome.
Change in Unified Parkinson's Disease Rating Scale section III (UPDRS III). | 36 weeks
  This scale can range from 0 to 132, and higher scores mean a worse outcome.
Change in Unified Parkinson's Disease Rating Scale section IV (UPDRS IV). | 36 weeks
  This scale can range from 0 to 24, and higher scores mean a worse outcome.
Change in objective assessment of gait measured by a sensor (MobilityLab) that assess step speed. | 36 weeks
Change in objective assessment of gait measured by a sensor (MobilityLab) that assess number of steps per minute. | 36 weeks
Change in objective assessment of gait measured by a sensor (MobilityLab) that assess distance between heels. | 36 weeks
Change in objective assessment of gait measured by a sensor (MobilityLab) that assess balance. | 36 weeks
Change in objective assessment of gait measured by Time Up and Go - Test 3 meters (TUG test 3M). | 36 weeks
Change in objective assessment of gait measured by Time Up and Go dual task - Test 3 meters (TUG dual task - test 3M). | 36 weeks
Change in objective assessment of gait measured by freezing of gait score (FOG score). | 36 weeks
Change in New Freezing of Gait Questionnaire (N-FOG). | 36 weeks
  This questionnaire can range from 0 to 28, and higher scores mean a worse outcome.
Change in Falls Efficacy Scale International (FES-I). | 36 weeks
  This questionnaire can range from 0 to 64, and higher scores mean a worse outcome.
Change in Activities-Specific Balance Confidence Scale (ABC scale). | 36 weeks
  This scale can range from 0 to 100%, and higher scores mean a better outcome.
Change in Beck Depression Inventory (BDI). | 36 weeks
  This inventory can range from 0 to 63, and higher scores mean a worse outcome.
Change in Beck Anxiety Inventory (BAI). | 36 weeks
  This inventory can range from 0 to 63, and higher scores mean a worse outcome.
Change in Starkstein Apathy Scale. | 36 weeks
  This scale can range from 0 to 42, and higher scores mean a worse outcome.
Change in Neuropsychiatric Inventory (NPI). | 36 weeks
Change in Ardouin Scale of Behavior in Parkinson's Disease. | 36 weeks
  This scale can range from 0 to 84, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo General Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gratwicke J, Zrinzo L, Kahan J, Peters A, Beigi M, Akram H, Hyam J, Oswal A, Day B, Mancini L, Thornton J, Yousry T, Limousin P, Hariz M, Jahanshahi M, Foltynie T. Bilateral Deep Brain Stimulation of the Nucleus Basalis of Meynert for Parkinson Disease Dementia: A Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):169-178. doi: 10.1001/jamaneurol.2017.3762. PMID 29255885
- [Result] Nombela C, Lozano A, Villanueva C, Barcia JA. Simultaneous Stimulation of the Globus Pallidus Interna and the Nucleus Basalis of Meynert in the Parkinson-Dementia Syndrome. Dement Geriatr Cogn Disord. 2019;47(1-2):19-28. doi: 10.1159/000493094. Epub 2019 Jan 10. PMID 30630160
- [Result] Sankar T, Lipsman N, Lozano AM. Deep brain stimulation for disorders of memory and cognition. Neurotherapeutics. 2014 Jul;11(3):527-34. doi: 10.1007/s13311-014-0275-0. PMID 24777384
- [Result] Kuhn J, Hardenacke K, Lenartz D, Gruendler T, Ullsperger M, Bartsch C, Mai JK, Zilles K, Bauer A, Matusch A, Schulz RJ, Noreik M, Buhrle CP, Maintz D, Woopen C, Haussermann P, Hellmich M, Klosterkotter J, Wiltfang J, Maarouf M, Freund HJ, Sturm V. Deep brain stimulation of the nucleus basalis of Meynert in Alzheimer's dementia. Mol Psychiatry. 2015 Mar;20(3):353-60. doi: 10.1038/mp.2014.32. Epub 2014 May 6. PMID 24798585
- [Result] Freund HJ, Kuhn J, Lenartz D, Mai JK, Schnell T, Klosterkoetter J, Sturm V. Cognitive functions in a patient with Parkinson-dementia syndrome undergoing deep brain stimulation. Arch Neurol. 2009 Jun;66(6):781-5. doi: 10.1001/archneurol.2009.102. PMID 19506141
- [Result] Wilson J, Yarnall AJ, Craig CE, Galna B, Lord S, Morris R, Lawson RA, Alcock L, Duncan GW, Khoo TK, O'Brien JT, Burn DJ, Taylor JP, Ray NJ, Rochester L. Cholinergic Basal Forebrain Volumes Predict Gait Decline in Parkinson's Disease. Mov Disord. 2021 Mar;36(3):611-621. doi: 10.1002/mds.28453. Epub 2020 Dec 31. PMID 33382126
- [Result] Muller ML, Bohnen NI. Cholinergic dysfunction in Parkinson's disease. Curr Neurol Neurosci Rep. 2013 Sep;13(9):377. doi: 10.1007/s11910-013-0377-9. PMID 23943367
- [Result] Gratwicke J, Zrinzo L, Kahan J, Peters A, Brechany U, McNichol A, Beigi M, Akram H, Hyam J, Oswal A, Day B, Mancini L, Thornton J, Yousry T, Crutch SJ, Taylor JP, McKeith I, Rochester L, Schott JM, Limousin P, Burn D, Rossor MN, Hariz M, Jahanshahi M, Foltynie T. Bilateral nucleus basalis of Meynert deep brain stimulation for dementia with Lewy bodies: A randomised clinical trial. Brain Stimul. 2020 Jul-Aug;13(4):1031-1039. doi: 10.1016/j.brs.2020.04.010. Epub 2020 Apr 22. PMID 32334074
- [Result] Dalrymple WA, Huss DS, Blair J, Flanigan JL, Patrie J, Sperling SA, Shah BB, Harrison MB, Druzgal TJ, Barrett MJ. Cholinergic nucleus 4 atrophy and gait impairment in Parkinson's disease. J Neurol. 2021 Jan;268(1):95-101. doi: 10.1007/s00415-020-10111-2. Epub 2020 Jul 28. PMID 32725313
- [Result] Koulousakis P, Andrade P, Visser-Vandewalle V, Sesia T. The Nucleus Basalis of Meynert and Its Role in Deep Brain Stimulation for Cognitive Disorders: A Historical Perspective. J Alzheimers Dis. 2019;69(4):905-919. doi: 10.3233/JAD-180133. PMID 31104014